CLINICAL TRIAL: NCT05321693
Title: Neuromodulatory Effects of Transcranial Pulsed Current Stimulation in Fibromyalgia: a Randomized Clinical Trial, Double-blinded, Controlled With Sham
Brief Title: Neuromodulatory Effects of Transcranial Pulsed Current Stimulation in Fibromyalgia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Andressa de Souza, Principal Investigador, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 49683221.2.0000.5307
Record Dates: First submitted 2022-03-25; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, double-blinded, parallel-group, sham-controlled trial to evaluate the superiority of tPCS in pain reduction in women with FM
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Based on the nature of the intervention, participants and physicians (health care providers/investigators) shall be blinded. Only one investigator will have access to the randomization list and will program the stimulation according to the list. The device comes programmed to perform the task input by the investigator, which will be trained by previous enrollment to the study onhow to perform the intervention. Sham stimulation occurs only for the initial 30seconds, afterwhich the patient should feelthat the body adjusts to the stimuli.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tPCS (Active Comparator)
  Interventions: Device: Transcranial Pulsed Current Stimulation
- Sham tPCS (Sham Comparator): The currentwill only be applied forthe first 30 seconds. Patients may notice the same sensation of initial stimulation butwill not receive the current for the remaining time.
  Interventions: Device: Transcranial Pulsed Current Stimulation

INTERVENTIONS:
Device: Transcranial Pulsed Current Stimulation — Current has a peak pulse amplitude of 2mA, with a frequency range from 6 to 10 Hz. A battery-powered current stimulator will be used. This device provides stimulation through biphasic and alternating square wave pulse, with random pulse width range from 1 to 20 ms

SUMMARY:
Fibromyalgia (FM) is a functional syndrome characterized by musculoskeletal, diffuse and persistent (> 3 months) chronic pain, that is also characterized by sleep disturbances, fatigue, humor changes and cognitive and psychological changes. Transcranial Pulsed Current Stimulation (tPCS) is a new Transcranial Electrical Stimulation (tES) that has been studied as a treatment option for chronic pain and neurological conditions . Studies have shown that tPCS is capable of pain and cognitive modulation; however, there are not enough studies with evidenceofits efficacy.Therefore, the primary aim of this study is to evaluate the effects of tPCS in pain, evaluated through Visual Analogue Scale (VAS) in FM patients; besides that, it is aimed to evaluate the effects of tPCS on quality of life, cognitive impairments, pain pressure threshold, descending inhibitory system of pain, and serum levels of Brain Derived Neurotrophic Factor (BDNF) and S100 Calcium-Binding Protein B (S100B). A randomized, double-blinded, controlled with sham clinical trial will be conducted with 70 (Critical f: 2.003; ES: 0.76; alpha: 0.05; power: 0.80) women with Fibromyalgia, from 30 to 65 years with pain on the Visual Analogue Scale (VAS) higher than 6 in the last 3 months. All patients will read and sign an Informed Consent Form (ICF). Each patient will be randomized to either 1+4 sessions of tPCS (2mA, 6-10Hz, 1-20ms, 20-25 minutes) or Sham. Patients will complete the following questionnaires/tests: Visual Analogue Scale (VAS), Pittsburgh Sleep Quality Index (PSQI), Fibromyalgia Impact Questionnaire (FIQ), Pain Catastrophizing Scale (PCS), Profile of Chronic Pain (PCP), Conditioned Pain Modulation Task (CPM-T), Pain Pressure Threshold Task (PPT-T), ReyAuditory-Verbal Learning Test (RAVLT), Controlled Oral Word Association Test (COWAT) and blood collection for serum levels of BDNF and S100B. For the main outcome, comparison between variables during time will be made through linear regression, with an adjustment for baseline levels and possible confounders.

DETAILED DESCRIPTION:
Recruitment: The study will be held in a clinical center at Novo Hamburgo (RS) -Brazil.Data collection will begin in December 2021, and it will end when sample size is achieved. A targeted approach will be used: recruiting referrals from clinics in the region of the study setting, along with patients from the clinical center where the trial will be conducted. Besides that, posters will be placed in common areas and posted on social media. Inclusion Criteria: women from 30 to 65 years old; FM diagnosis according to ACR criteria (2016); pain on VAS equal to or higher than 6 in the last 3 months; chronic stable treatment over the past 3 months.

Exclusion Criteria: pregnancy or lack of contraceptive use; history of alcohol or drug abuse in the last 6 months, neurological disorders, cardiac arrhythmia; use of drugs that change vascular response; history of head trauma, mild or severe, neurosurgery; decompensated systemic diseases; current diagnosis or history of cancer.

tPCSThe procedure will begin with placement of bilateral circular electrodes in the inferior ear lobe (ECG position A1) fixed by an ear clip. The electrode's radius will be approximately 0.785cm2. Current has a peak pulse amplitude of 2mA, with a frequency range from 6 to 10 Hz. A battery-powered current stimulator will be used. This device provides stimulation through biphasic and alternating square wave pulse, with random pulse width range from 1 to 20 ms. tPCS sessions will last 20 minutes plus 5 minutes for setting up, meanwhile when questionnaires and tests are applied, sessions can last 1 to 2 hours. Sessions will be made in a 1+4 way, in which outcomes will be evaluated before and after the first session and after the last session. Studies display evidence of clinical improvement after 5 sessions of transcranial electrical stimulation in FM. A standardized questionnaire will be performed in order to observe adverse effects immediately after the intervention.Sham tPCSThe current will only be applied for the first 30 seconds. Patients may notice the same sensation of initial stimulation but will not receive the current for the remaining time. Analogue to tPCS, 5 sessions will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Women from 30 to 65 years old
* FM diagnosis according to ACR criteria (2016)
* Pain on VAS equal to or higher than 6 in the last 3 months
* Chronic stable treatment over the past 3 months.

Exclusion Criteria:

* Pregnancy or lack of contraceptive use;
* History of alcohol or drug abuse in the last 6 months,
* Neurological disorders;
* Cardiac arrhythmia;
* Use of drugs that change vascular response;
* History of head trauma, mild or severe;
* History of neurosurgery;
* Decompensated systemic diseases;
* Current diagnosis or history of cancer

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
Pain on Visual Analogue Scale (VAS) | Change from day 5 to baseline
  a continuous scale from 0-100mm, considering 60mm as the minimum for chronic pain

SECONDARY OUTCOMES:
Quality of Sleep | Change from day 5 to baseline
  Pittsburgh Sleep Quality Index (PSQI) - from 0 to 21. The higher the worse
Impact of Fibromyalgia | Change from day 5 to baseline
  Fibromyalgia Impact Questionnaire (FIQ), subdivided into overall impact, symptoms and function. From 0 to 100. The higher the worse
Pain Catastrophizing | Change from day 5 to baseline
  Pain Catastrophizing Scale (PCS), subdivided into magnification, rumination, and hopelessness. From 0 to 52. The higher the worse
Profile of Pain | Change from day 5 to baseline
  Profile of Chronic Pain (PCP), subdivided into pain intensity and frequency (1-4), the impact of pain in activities (5-10), and impact of pain in emotions (11-15). The higher the worse
Descending Inhibitory System | Change from day 5 to baseline
  Conditioned Pain Modulation task: evaluate the descending inhibitory system of pain, measured by the difference of pain (VAS) between two painful stimuli. From -6 to 4. As far from 0 the worse
Pain Pressure Threshold | Change from day 5 to baseline
  anelectronic algometer will be placed in the forearm, patient will report first pain sensation and maximum pain. Starts in 0. The closer to zero the worst.
Serum levels of BDNF, S100B, and estradiol | Change from day 5 to baseline
  ELISA Technique. Starts in 0
Cognitive Impairment | Change from day 5 to baseline
  Controlled Oral Word Association Test (COWAT) for cognitive evaluation. Starts in 0. The higher the better

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Universidade La Salle, Canoas, Rio Grande do Sul
  - Instituto de Neuromodulação e Reabilitação Avançada, Novo Hamburgo, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No